CLINICAL TRIAL: NCT05675306
Title: Dose Frequency Randomized Control Trial for Dynamic Temporal and Tactile Cueing (DTTC) Treatment for Childhood Apraxia of Speech
Brief Title: Dose Frequency RCT on DTTC in Children With CAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Collaborators: Hofstra University (Other); New York University (Other); University of Vermont (Other); University of Sydney (Other); Remarkable Speech and Movement (Unknown)
Responsible Party: Principal Investigator, Jenya Iuzzini-Seigel, Assistant Professor, Marquette University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 75245
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Childhood Apraxia of Speech
Keywords: treatment; dose frequency; speech sound disorders; cumulative dosage; whole word accuracy; Dynamic Temporal and Tactile Cueing; DTTC; Childhood apraxia of speech
MeSH Terms: conditions — Apraxias; Speech Sound Disorder

STUDY DESIGN:
Intervention Model Description: The proposed work is multisite Phase III parallel-group RCT that aims to investigate the outcomes of DTTC in children with CAS and determine whether dose frequency impacts response to treatment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Dose Frequency (Experimental): This group will receive treatment 4x/week for 6 weeks
  Interventions: Behavioral: Dynamic Temporal and Tactile Cueing Treatment
- Low Dose Frequency (Active Comparator): This group will receive treatment 2x/week for 12 weeks
  Interventions: Behavioral: Dynamic Temporal and Tactile Cueing Treatment

INTERVENTIONS:
Behavioral: Dynamic Temporal and Tactile Cueing Treatment — DTTC is a dynamic, motor-based treatment approach designed for children with severe CAS. This approach is based on Integral Stimulation (Edeal & Gildersleeve-Neumann, 2011; Maas & Farinella, 2012; Maas et al., 2019; Strand & Debertine, 2000; Strand & Skinder, 1999), in which the clinician instructs the child to "listen to me, watch me, and do what I do" and systematically taxes and supports the speech motor system to facilitate system-wide change in speech output (Strand, 2020).
  Other Names: DTTC

SUMMARY:
Childhood apraxia of speech (CAS) is a pediatric motor-based speech sound disorder that requires a specialized approach to intervention (Maas et al., 2014). The extant literature on the treatment of CAS commonly recommends intensive treatment using a motor-based approach, with some of the best evidence supporting the use of Dynamic Temporal and Tactile Cueing (DTTC; Strand, 2020). To date, a rigorous and systematic comparison of high and low dose frequency has not been undertaken for DTTC, resulting in a lack of evidence to guide decisions about the optimal treatment schedule for this intervention. The current study aims to fill this gap in knowledge by comparing treatment outcomes when dose frequency is varied.

The goal of this clinical trial is to determine whether the number of treatment sessions per week has an effect on intervention outcomes in 60 children with CAS. The main question this research will address is whether whole word accuracy will differ between two groups of children undergoing DTTC treatment when one group of children receives treatment twice a week for 12 weeks and the other group receives treatment 4 times a week for 6 weeks. Community clinicians will administer all treatment sessions.

DETAILED DESCRIPTION:
Sixty children with childhood apraxia of speech will be treated with DTTC treatment. A Phase III randomized controlled trial with parallel groups will be conducted to compare effects of low versus high dose frequency on DTTC treatment outcomes in children with CAS. Children with CAS between 2;5-7;11 years of age will be recruited to participate in this study. Treatment will be provided in the community setting by speech-language pathologists who have completed specialized training administering DTTC in a research reliable manner.

True randomization with concealed allocation will be used to assign children to either the low or high dose frequency group. Treatment will be administered in 1-hour sessions either 4 times per week over a 6-week period (high dose) or 2 times per week over a 12-week period (low dose) for a total of 24 hours per child. To measure treatment gains, probe data will be collected before treatment, during treatment, and 1 day, 1 week, 4 weeks, and 12 weeks post-treatment. Probe data will consist of customized treated words and a standard set of untreated words to assess generalization of treatment gains. The primary outcome variable will be whole word accuracy, a measure of segmental, phonotactic, and suprasegmental accuracy.

This will be the first randomized controlled trial (RCT) to evaluate dose frequency for DTTC treatment in children with CAS.

ELIGIBILITY:
Inclusion Criteria:

1. CAS diagnosis confirmed by research team as described below (e.g., Iuzzini-Seigel et al., 2022; Shriberg et al., 2017; Strand & McCauley, 2019),
2. 2;6-7;11 years of age at treatment commencement;
3. English as the primary language;

Exclusion Criteria:

1. concomitant developmental disorders (including autism, global developmental delay, intellectual disability);
2. diagnosis of severe or primary dysarthria as described below;
3. palatal or structural orofacial anomalies as described below,
4. uncorrected vision impairment
5. hearing loss;
6. receiving speech treatment elsewhere over the course of this study, although language, augmentative and alternative communication treatment, or similar non-speech treatment, would be permitted
7. Receptive Language Index standard score less than 70 on the Receptive-Expressive Emergent Language Test, 4th edition (REEL-4; Brown et al., 2020) for children 2-3 years of age, the Clinical Evaluation of Language Fundamentals - Preschool 3rd edition (CELF-P3; Wiig et al., 2020) for children 4-5 years of age, or the Clinical Evaluation of Language Fundamentals - 5th edition (CELF-5; Wiig et al., 2013) for children 6-7 years of age,
8. Nonverbal Index standard score less than 70 on the Reynolds Intellectual Assessment Scales- 2nd edition, Remote (Reynolds & Kamphaus, 2015), and
9. no evidence of communicative intent, attempts at verbal communication, focused attention to the clinician's face, or demonstrated ability to imitate during the DEMSS.

Ages: 30 Months to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes to whole word accuracy | Pre to post-treatment follow-up (6-12 weeks of treatment plus 12 weeks post completion of treatment)
  A multi-factor whole word accuracy measure (Multilevel word Accuracy Composite Scale; Case et al., under review) that systematically accounts for segmental and prosodic accuracy, word shape maintenance, and smoothness and fluency of movement transitions will be calculated on treated and similar untreated words in the generalization probe.

SECONDARY OUTCOMES:
Phoneme accuracy | Pre to post-treatment follow-up (6-12 weeks of treatment plus 12 weeks post completion of treatment)
  Percentage of phonemes correct on the generalization probe
Speech Intelligibility | Pre to post-treatment follow-up (6-12 weeks of treatment plus 4 weeks post completion of treatment)
  Calculated based on the Intelligibility in Context Scale (McLeod et al., 2012), a parent survey measure
Functional communication | Pre to post-treatment follow-up (6-12 weeks of treatment plus 4 weeks post treatment)
  Calculated based on the Functional Outcomes on Communication Under Six (Thomas-Stonell et al., 2015), a parent survey measure

CONTACTS AND LOCATIONS:
Overall Officials: Jenya Iuzzini-Seigel, PhD, Principal Investigator — Marquette University
Locations (1):
- Marquette U, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual level data will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months after publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal and evidence of ethical conduct of research and appropriate institutional oversight (e.g., IRB). Proposals should be directed to jenya.iuzzini-seigel@marquette.edu. To gain access, data requestors will need to complete and sign a data sharing agreement.

REFERENCES:
- [Background] Wiig, E. H., Secord, W. A., & Semel, E. M. (2020). Clinical Evaluation of Language Fundamentals - Preschool (3rd ed.). Pearson.
- [Result] Strand EA. Dynamic Temporal and Tactile Cueing: A Treatment Strategy for Childhood Apraxia of Speech. Am J Speech Lang Pathol. 2020 Feb 7;29(1):30-48. doi: 10.1044/2019_AJSLP-19-0005. Epub 2019 Dec 17. PMID 31846588
- [Result] Maas E, Gildersleeve-Neumann C, Jakielski KJ, Stoeckel R. Motor-based intervention protocols in treatment of childhood apraxia of speech (CAS). Curr Dev Disord Rep. 2014 Sep;1(3):197-206. doi: 10.1007/s40474-014-0016-4. PMID 25313348
- [Result] Edeal DM, Gildersleeve-Neumann CE. The importance of production frequency in therapy for childhood apraxia of speech. Am J Speech Lang Pathol. 2011 May;20(2):95-110. doi: 10.1044/1058-0360(2011/09-0005). Epub 2011 Feb 17. PMID 21330650
- [Result] Maas E, Farinella KA. Random versus blocked practice in treatment for childhood apraxia of speech. J Speech Lang Hear Res. 2012 Apr;55(2):561-78. doi: 10.1044/1092-4388(2011/11-0120). Epub 2011 Dec 29. PMID 22207698
- [Result] Maas E, Gildersleeve-Neumann C, Jakielski K, Kovacs N, Stoeckel R, Vradelis H, Welsh M. Bang for Your Buck: A Single-Case Experimental Design Study of Practice Amount and Distribution in Treatment for Childhood Apraxia of Speech. J Speech Lang Hear Res. 2019 Sep 20;62(9):3160-3182. doi: 10.1044/2019_JSLHR-S-18-0212. Epub 2019 Aug 19. PMID 31425660
- [Result] Iuzzini-Seigel J, Allison KM, Stoeckel R. A Tool for Differential Diagnosis of Childhood Apraxia of Speech and Dysarthria in Children: A Tutorial. Lang Speech Hear Serv Sch. 2022 Oct 6;53(4):926-946. doi: 10.1044/2022_LSHSS-21-00164. Epub 2022 May 6. PMID 35523425
- [Result] Shriberg LD, Strand EA, Fourakis M, Jakielski KJ, Hall SD, Karlsson HB, Mabie HL, McSweeny JL, Tilkens CM, Wilson DL. A Diagnostic Marker to Discriminate Childhood Apraxia of Speech From Speech Delay: Introduction. J Speech Lang Hear Res. 2017 Apr 14;60(4):S1094-S1095. doi: 10.1044/2016_JSLHR-S-16-0148. PMID 28384695
- [Result] Goldman, R., & Fristoe, M. (2015). Goldman-Fristoe Test of Articulation - Third Edition (GFTA-3). Pearson Assessments.
- [Result] Strand, E. A., & Debertine, P. (2000). The efficacy of integral stimulation intervention with developmental apraxia of speech. Journal of Medical Speech-Language Pathology, 8(4), 295-300.
- [Result] Strand, E. A., & McCauley, R. J. (2019). The Dynamic Evaluation of Motor Speech Skill (DEMSS). Brookes.
- [Result] Thomas-Stonell, N., Oddson, B., Robertson, B., Walker, J. & Rosenbaum, P. (2015). The FOCUS©-34: Focus on the Outcomes of Communication Under Six. Holland Bloorview Kids Rehabilitation Hospital, Toronto, ON. http://www.focusoutcomemeasurement.ca
- [Result] Wiig, E. H., Semel, E. M., & Secord, W. A. (2013). Clinical Evaluation of Language Fundamentals - 5. Pearson.
- [Derived] Iuzzini-Seigel J, Case J, Grigos MI, Velleman SL, Thomas D, Murray E. Dose frequency randomized controlled trial for Dynamic Temporal and Tactile Cueing (DTTC) treatment for childhood apraxia of speech: protocol paper. BMC Pediatr. 2023 May 25;23(1):263. doi: 10.1186/s12887-023-04066-2. PMID 37226208